CLINICAL TRIAL: NCT03776786
Title: Phase 1 First-in-Human, Time Lagged, Single Ascending Dose Study of TY014 in Healthy Adult Volunteers (Safety Arm - 1A) and Sequential Time Lagged, Parallel-Group, Randomised, Placebo-Controlled, Double-Blind, Single Ascending Dose Study of TY014 in YF-17D Vaccine Strain-Challenged Healthy Adult Volunteers (Efficacy Arm - 1B)
Brief Title: Safety and Tolerability of an Antibody Against Yellow Fever Virus (TY014) in Humans
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Tysana Pte Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YFT-001; CTA1800118 (Other: Health Sciences Authority of Singapore)
Record Dates: First submitted 2018-12-12; First posted 2018-12-17 (Actual); Last update posted 2019-10-25 (Actual); Status verified 2019-10

CONDITIONS: Treatment of Acute Yellow Fever Virus Infection
MeSH Terms: interventions — TY014; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (14):
- Safety Arm - 0.5 mg/kg (Experimental): Subject will be administered with 0.5 mg/kg of TY014 via IV infusion over a period of 30 minutes.
  Interventions: Biological: TY014
- Safety Arm - Placebo (Placebo Comparator): Subject will be administered with 0.9% saline via IV infusion over a period of 30 minutes.
  Interventions: Other: 0.9% Saline
- Safety Arm - 2 mg/kg (Experimental): Subject will be administered with 2 mg/kg of TY014 via IV infusion over a period of 30 minutes.
  Interventions: Biological: TY014
- Safety Arm - 5 mg/kg (Experimental): Subject will be administered with 5 mg/kg of TY014 via IV infusion over a period of 30 minutes.
  Interventions: Biological: TY014
- Safety Arm - 10 mg/kg (Experimental): Subject will be administered with 10 mg/kg of TY014 via IV infusion over a period of 30 minutes.
  Interventions: Biological: TY014
- Safety Arm - 20 mg/kg (Experimental): Subject will be administered with 20 mg/kg of TY014 via IV infusion over a period of 30 minutes.
  Interventions: Biological: TY014
- Efficacy Arm - 2 mg/kg (Experimental): Subject will be administered with 2 mg/kg of TY014 via IV infusion over a period of 30 minutes 24 hours post-YF vaccination.
  Interventions: Biological: TY014
- Efficacy Arm - 2 mg/kg Placebo (Placebo Comparator): Subject will be administered with 0.9% saline via IV infusion over a period of 30 minutes 24 hours post-YF vaccination.
  Interventions: Other: 0.9% Saline
- Efficacy Arm - 5 mg/kg (Experimental): Subject will be administered with 5 mg/kg of TY014 via IV infusion over a period of 30 minutes 24 hours post-YF vaccination.
  Interventions: Biological: TY014
- Efficacy Arm - 5 mg/kg Placebo (Placebo Comparator): Subject will be administered with 0.9% saline via IV infusion over a period of 30 minutes 24 hours post-YF vaccination.
  Interventions: Other: 0.9% Saline
- Efficacy Arm - 10 mg/kg (Experimental): Subject will be administered with 10 mg/kg of TY014 via IV infusion over a period of 30 minutes 24 hours post-YF vaccination.
  Interventions: Biological: TY014
- Efficacy Arm - 10 mg/kg Placebo (Placebo Comparator): Subject will be administered with 0.9% saline via IV infusion over a period of 30 minutes 24 hours post-YF vaccination.
  Interventions: Other: 0.9% Saline
- Efficacy Arm - 20 mg/kg (Experimental): Subject will be administered with 20 mg/kg of TY014 via IV infusion over a period of 30 minutes 24 hours post-YF vaccination.
  Interventions: Biological: TY014
- Efficacy Arm - 20 mg/kg Placebo (Placebo Comparator): Subject will be administered with 0.9% saline via IV infusion over a period of 30 minutes 24 hours post-YF vaccination.
  Interventions: Other: 0.9% Saline

INTERVENTIONS:
Biological: TY014 — TY014 Injection, (100 mg/5 mL/Vial), Yellow Fever Virus (YFV) Monoclonal Antibody (mAb)
  Arms: Efficacy Arm - 10 mg/kg; Efficacy Arm - 2 mg/kg; Efficacy Arm - 20 mg/kg; Efficacy Arm - 5 mg/kg; Safety Arm - 0.5 mg/kg; Safety Arm - 10 mg/kg; Safety Arm - 2 mg/kg; Safety Arm - 20 mg/kg; Safety Arm - 5 mg/kg
Other: 0.9% Saline — Placebo
  Arms: Efficacy Arm - 10 mg/kg Placebo; Efficacy Arm - 2 mg/kg Placebo; Efficacy Arm - 20 mg/kg Placebo; Efficacy Arm - 5 mg/kg Placebo; Safety Arm - Placebo

SUMMARY:
Yellow Fever is an acute viral hemorrhagic disease caused by the Yellow Fever Virus (YFV), a re-emerging arbovirus transmitted by the same mosquito vector (Aedes aegypti) that transmits Dengue virus (DENV) and Zika virus (ZIKV). YFV is endemic in tropical and subtropical areas of South America and Africa, causing an estimated 200,000 infections and 30,000 deaths annually. It has now become a growing public health problem, rapidly spreading throughout the two (2) continents in a cyclical pattern. With climate change, global travel and urbanisation, which increase the chance for mosquito-borne diseases to spread rapidly, the risk of YFV establishing its foothold in the Asia-Pacific region with periodic epidemic bursts remains a real public health concern.

Although there is currently a safe and effective vaccine available on the market, global shortages of supplies have severely hampered any efforts in the prevention and control of YFV outbreaks. To date, no YFV therapy (biologic or small molecule) has advanced to clinical trials. TY014 will be the first therapeutic in the world, specifically targeting YFV, to enter clinical trials. It is anticipated that a monoclonal antibody therapeutic could be administered to infected cases to reduce disease severity within the patient and their contacts.

This is a Phase 1, first-in-human TY014, YFV monoclonal antibody (mAb), study to be conducted in two (2) arms:

* Safety Arm (1A): Healthy adult volunteers
* Efficacy Arm (1B): Healthy adult volunteers challenged with YF-17D Vaccine Strain 24 hours prior to TY014 dosing

TY014 will be administered once through single IV infusion over 30 minutes. Total duration of study participation is estimated at approximately 114 days from the date of screening.

The main objectives of this study are to: (a) evaluate the safety of TY014 in healthy adult volunteers, and (b) evaluate the safety of TY014 in YF-17D Vaccine Strain-challenged healthy adult volunteers. Percentage aviremia of YF-17D Vaccine Strain-challenged subjects within 48 hours after IV infusion of TY014 will also be assessed.

DETAILED DESCRIPTION:
Safety Arm (1A):

Safety Arm is a phase 1A First-in-Human, Time Lagged, Single Ascending Dose Study of TY014 in Healthy Adult Volunteers.

Safety, tolerability and PK of TY014 will be assessed. The dose escalation will include 27 healthy volunteers in five (5) dose cohorts:

* 0.5 mg/kg, N = 2 TY014 + 5 Placebos
* 2 mg/kg, N = 5 TY014
* 5 mg/kg, N = 5 TY014
* 10 mg/kg, N = 5 TY014
* 20 mg/kg, N = 5 TY014 Subjects will be required to be inpatient at the trial site for approximately 72 hours.

Dose escalations will be guided by a safety review of clinical signs, adverse events (AEs), and laboratory tests (excluding lipase) of the prior group (up to 48 hours post-dose for cohort 1, and up to Day 7 post-dose for cohorts 2 - 5).

A minimum of 20-hour interval from the first TY014 treatment subject dosing must take place before the second TY014 treatment subject can be dosed within each cohort. No such time interval will be required for dosing of subsequent TY014 treatment subjects (third subject onwards) within the same cohort, as well as Placebo dosing in dose cohort 1 (i.e. all five placebos can be dosed at the same time).

After 72 hours, subjects will be discharged from trial site and to return for scheduled follow-up visits.

Subjects will be followed for up to approximately Day 84 for PK sampling, with serum samples taken at specified times.

Dose escalations for the Safety (1A) Arm will be guided by a safety review of clinical signs, adverse events (AEs), and laboratory tests (excluding lipase) of the prior dose cohort (up to Day 7).

Similar safety review (up to Day 7) will also be completed for the equivalent dose in Safety Arm (1A) prior to the commencement of the Efficacy Arm (1B) for each specified dose.

Efficacy Arm (1B):

Efficacy Arm is a phase 1B Sequential Time Lagged, Parallel-Group, Randomised, Placebo-Controlled, Double-Blind, Single Ascending Dose Study of TY014 in YF-17D Vaccine Strain-Challenged Healthy Adult Volunteers.

Safety, tolerability and time to achieve aviremia through negative YFV isolation from blood in YF-17D Vaccine Strain-challenged healthy adult volunteers when given an IV infusion of TY014 will be assessed.

Eligible subjects will be randomised into TY014 or Placebo Group in each cohort.

The dose escalation will include up to 40 healthy volunteers in up to four (4) dose cohorts:

* 2 mg/kg, N = 5 TY014 + 5 Placebos
* 5 mg/kg, N = 5 TY014 + 5 Placebos
* 10 mg/kg, N = 5 TY014 + 5 Placebos
* 20 mg/kg, N = 5 TY014 + 5 Placebos Efficacy Arm (1B) will be based on an adaptive trial design, with ten (10) YF-17D vaccinated subjects from each dose cohort being randomised 1:1 into either TY014 or Placebo group, five (5) subjects in each group. After TY014 or placebo administration, safety and efficacy of TY014 in YF-17D Vaccine Strain-Challenged subjects will be assessed.

  i) If current dose of TY014 shows safety but not efficacy*, Efficacy Arm (1B) will escalate to the next dose cohort.

ii) If current dose of TY014 is safe and efficacious*, efficacious dose of TY014 is established and the Efficacy Arm (1B) of the trial is completed.

*Efficacy of TY014 is defined as aviremia by virus isolation being observed in 100% of vaccinated subjects within 48 hours post-dosing.

Subjects will be required to be inpatient at the trial site for approximately 96 hours.

Subjects will be vaccinated with the YF-17D Vaccine on Day -1. On Day 0, 24 hours after vaccination, subjects will then be administered TY014 or Placebo.

A minimum of 20-hour interval from the first two (2) subjects dosing (1 treatment and 1 placebo concurrently) must take place before the third subject can be dosed within each cohort. No such time interval will be required for dosing of subsequent subjects (fourth subject onwards) within the same cohort.

After 96 hours, subjects will be discharged from trial site and are to return for scheduled follow-up visits.

PD and PK measurements will be conducted at various time points throughout the study. Subjects will be followed for up to approximately Day 84 post-dose. Samples for PD (serum and urine) and PK (serum) assessments will be taken at specified time points.

Dose escalations for the Efficacy (1B) Arm will be guided by a safety review of clinical signs, adverse events (AEs), laboratory tests (excluding lipase) and presence of viremia (via virus isolation) of the prior dose cohort (up to Day 14). Escalation to the next dose cohort (e.g. from dose cohort 1 (2 mg/kg) to dose cohort 2 (5 mg/kg), from dose cohort 2 (5 mg/kg) to dose cohort 3 (10 mg/kg) and from dose cohort 3 (10 mg/kg) to dose cohort 4 (20 mg/kg)) will only be conducted if from prior dose cohort (e.g. dose cohort 1 (2 mg/kg), dose cohort 2 (5 mg/kg) and dose cohort 3 (10 mg/kg) respectively):

1. safety (up to Day 14 post-dose) has been established through a safety review, and
2. presence of viremia (up to 48 hours post-dose) via virus isolation in any of the TY014-treated subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult volunteers, aged 21 to 50 years old, men or women
2. Subjects negative for human immunodeficiency virus (HIV), Hepatitis B virus surface Antigen (HBsAg) and Hepatitis C virus (HCV)
3. Subjects who have not been vaccinated against or had prior exposure to Yellow Fever Virus (YFV)
4. Subjects who have no history of travels to Central America, South America, Africa or any other YF endemic countries, and have no plans to visit Central America, South America, Africa or any other YF endemic countries in the next six (6) months
5. Subjects who are willing to comply with the requirements of the study protocol, attend scheduled visits and make themselves available for the duration of the study with access to a consistent means of telephone contact, which may be, but not limited to, at home or at work via landline or mobile
6. Subjects who give written informed consent approved by the Ethical Review Board governing the site
7. Satisfactory baseline medical assessment as assessed by physical examination and a stable health status. Normal laboratory values must be within normal range of the assessing site or show minor variations that are deemed not clinically significant as judged by the Investigator and acceptable for study entry. A stable health status is defined as the absence of a health event satisfying the definition of a serious adverse event
8. Accessible vein in the forearm for blood collection
9. Female subjects of childbearing potential may be enrolled in the study if they have negative urine pregnancy tests on the day of screening and day of admission
10. Female subjects of non-childbearing potential due to surgical sterilization (hysterectomy or bilateral oophorectomy or tubal ligation) or menopause. Post-menopause subjects must have had at least 12 months of natural (spontaneous) amenorrhea
11. Both male (if he has a partner of childbearing potential) and female subjects (of childbearing potential) must agree to use adequate and reliable contraceptive measures (e.g. spermicides, condoms, contraceptive pills, etc.) or practice abstinence throughout the duration of the study (up to 84 days post-dosing)

Exclusion Criteria:

1. Presence of acute infection in the preceding 14 days, or presence of a temperature ≥ 38.0 ˚C (oral or tympanic temperature assessment), or acute symptoms greater than of "mild" severity on the scheduled date of admission
2. History of severe drug and / or food allergies and / or known allergies to the trial product or its components
3. Female subject who is pregnant or breast-feeding
4. History or presence of cardiovascular, respiratory, hepatic, renal, gastrointestinal, neuropsychiatric, or immunosuppressive disorders
5. Evidence of clinically significant anaemia (HB < 10 g/dL) or any other significant active haematological disease, or having donated > 450 mL of blood within the past three (3) months
6. Evidence of substance abuse, or previous substance abuse
7. Participation or planned participation in a study involving the administration of an investigational compound within the past four (4) months or during this study period
8. Receipt of immunoglobulins and/or any blood products within nine (9) months of study enrolment or planned administration of any of these products during the study period
9. Administration of any licensed vaccine within 30 days before the first study vaccine dose.
10. History of any reaction to monoclonal antibodies
11. Any condition that, in the opinion of the Investigator, would complicate or compromise the study or well-being of the subject
12. Both male (if he has a partner of childbearing potential) and female subjects (of childbearing potential) who are unwilling to use adequate contraception or practice abstinence throughout the duration of the study (up to 84 days post-dosing)

Efficacy Arm (1B) only:

Subjects meeting any of the following criteria will be excluded from the study:

1. Planned travels to Central America, South America, Africa or any other YFV-endemic countries in the next six (6) months
2. History of thymus gland disease.
3. Diagnosed with cancer or on treatment for cancer with the three (3) years prior to the screening.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2018-12-06 (Actual); Primary Completion 2019-07-01 (Actual); Study Completion 2019-10-10 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Event (Safety and Tolerability) | 84 Days
  Presence or absence of infusion reaction (hypersensitivity / anaphylaxis / etc.) in dose cohorts.
Percentage Aviremia Post Treatment (Efficacy Arm only) | 14 Days
  Percentage of YF-17D Vaccine Strain-challenged healthy adult volunteers showing aviremia via virus isolation within 48 hours after given an IV infusion of TY014

SECONDARY OUTCOMES:
Maximum Concentration (Cmax) - Pharmacokinetic Assessment | 84 Days
  Constant monitoring of the levels of antibody in subject sera through various time points as stated below would help elucidate the maximum concentration (Cmax) of TY014 in human serum.
Time to Maximum Concentration (Tmax) - Pharmacokinetic Assessment | 84 Days
  Constant monitoring of the levels of antibody in subject sera through various time points as stated below would help elucidate the time to maximum concentration (Tmax) of TY014 in human serum.
Area Under the Curve Extrapolated to Infinity (AUC0-∞) - Pharmacokinetic Assessment | 84 Days
  Constant monitoring of the levels of antibody in subject sera through various time points as stated below would help elucidate the area under the curve extrapolated to infinity (AUC0-∞) of TY014.
AUC calculated from time of administration to the last measurable concentration (AUC0-last) - Pharmacokinetic Assessment | 84 Days
  Constant monitoring of the levels of antibody in subject sera through various time points as stated below would help elucidate the AUC calculated from time of administration to the last measurable concentration (AUC0-last) of TY014.
Half-Life (t1/2) - Pharmacokinetic Assessment | 84 Days
  Constant monitoring of the levels of antibody in subject sera through various time points as stated below would help elucidate the half-life (t1/2) of TY014 in human serum.
Volume of Distribution (Vd) - Pharmacokinetic Assessment | 84 Days
  Constant monitoring of the levels of antibody in subject sera through various time points as stated below would help elucidate the volume of distribution (Vd) of TY014 in human serum.
Clearance [CL] - Pharmacokinetic Assessment | 84 Days
  Constant monitoring of the levels of antibody in subject sera through various time points as stated below would help elucidate clearance [CL] of TY014 in human serum.
Viral Load Reduction (Efficacy Arm only) | 84 Days
  Assess YFV viral load reduction from blood by quantitative reverse transcriptase-polymerase chain reaction (qRT-PCR) in YF-17D Vaccine Strain-challenged healthy adult volunteers when given an IV infusion of TY014.

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Low, MBBS, Principal Investigator — Singapore General Hospital
Locations (1):
- SingHealth Investigational Medicine Unit, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Low JG, Ng JHJ, Ong EZ, Kalimuddin S, Wijaya L, Chan YFZ, Ng DHL, Tan HC, Baglody A, Chionh YH, Lee DCP, Budigi Y, Sasisekharan R, Ooi EE. Phase 1 Trial of a Therapeutic Anti-Yellow Fever Virus Human Antibody. N Engl J Med. 2020 Jul 30;383(5):452-459. doi: 10.1056/NEJMoa2000226. PMID 32726531